CLINICAL TRIAL: NCT01282697
Title: Phase I Clinical Trial of Rapamycin and Irinotecan in Pediatric Patients With Refractory Solid Tumors
Brief Title: Clinical Trial of Rapamycin and Irinotecan in Pediatric Patients With Refractory Solid Tumors
Acronym: RAPIRI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4791
Record Dates: First submitted 2010-11-12; First posted 2011-01-25 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Refractory Solid Tumors in Children
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rapamycin+irinotecan at a given dose (Experimental)
  Interventions: Drug: Combined administration of irinotecan and rapamycin

INTERVENTIONS:
Drug: Combined administration of irinotecan and rapamycin — This phase I trial is a dose escalation study of irinotecan + rapamycin with a 3+3 statistical design.

SUMMARY:
Therapeutic solutions to treat solid tumors that are resistant to conventional treatments are now limited. Laboratory data in animals (on pediatric tumors such as brain tumors, sarcomas and neuroblastomas) have shown that the combination of irinotecan (HIF1alpha inhibitor) and rapamycin (mTOR inhibitor) allowed to block development of blood vessels in the tumor and could, in some cases, stop its progression. This drug combination has already been tested in adult patients with refractory tumors and seems to give encouraging results with stabilization of the tumor. The dose and toxicity of irinotecan and rapamycin are known when these drugs are administered separately and in a context different from that of refractory tumors. RAPIRI is a phase I clinical trial whose principal objectives are to determine the maximum dose at which these two molecules may be administered and to assess the safety of this new combination of drugs.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 1 year old and =< 21 years old;
* Refractory solid tumors, histologically proven at diagnosis (no additional biopsy needs to be performed for the purpose of the study);
* Relapsed or refractory solid tumors after standard treatment or phase II, III-IV clinical trials treatment have failed;
* Karnofsky or Lansky status >= 70%;
* Life expectancy >= 8 weeks;
* No chemotherapy / radiotherapy within 4 weeks before entry into the study;
* Adequate biological parameters :

  * Absolute neutrophil count >= 1.0 x 109/L;
  * Platelet count >= 100 x 109/L;
  * Hemoglobin >= 8 mg/dL;
  * Total bilirubine =< 1.5 ULN;
  * Transaminases =< 2.5 ULN (=< 5 ULN in case of liver metastases);
  * Creatinine clearance (Cockroft) >= 70 mL/min/1.73 m2;
  * Normal coagulation profile with prothrombin >= 70%, TCA =< 35 and fibrinogen >= 2 g/L;
* Patients with 1 to 3 previous therapeutic lines are eligible;
* No current grade >= 2 organ toxicity based on NCI-CTCAE version 3.0;
* All patients with reproductive potential must have an effective method of birth control while on study;
* Negative pregnancy test in females when indicated;
* Informed written consent signed by patients or their parents or legal guardians;
* Patient who was informed of the results of prior medical consultation;
* Patient having a social insurance.

Exclusion Criteria:

* Patient with a constitutional anomaly of coagulation and/or of hemostasis (type hemophilia, von Willebrand disease, congenital clotting factor deficit, platelet disorder), exposing them to increased risk of bleeding;
* Pre-treatment with a mTOR inhibitor;
* Other simultaneous malignancy;
* Concurrent administration of any other anti-tumour therapy;
* Known hypersensitivity or contraindication to study drugs or ingredients;
* Severe concomitant disease (e.g. infection disease);
* Patient unable for medical follow-up;
* Pregnancy and/or lactation;
* Patient included in another clinical drug trial;
* Patient taking drugs interfering with pharmacology of rapamycin and/or irinotecan (e.g. drugs interfering with CYP3A4);
* Patient under judicial protection.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2011-04-22 (Actual); Primary Completion 2013-02-20 (Actual); Study Completion 2013-02-20 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) of irinotecan and rapamycin combination in children with refractory solid tumors. | 28 days
  The Dose-Limiting Toxicity (DLT) of the drug combination is determined during the first cycle (J1 to J28) of treatment. MTD will be defined as the dose level immediately below the dose level at which 2 patients in a cohort of 3 to 6 patients will have experienced a DLT.
Characterize the pharmacokinetics of rapamycin and irinotecan during the first cycle of treatment. | Day1 + day8
  Pharmacokinetic parameters for rapamycin will be evaluated at days 1 and 8 of the first cycle of treatment. Pharmacokinetic parameters for irinotecan will be evaluated at day 1 of the first cycle of treatment. Pharmacokinetic profile will be modelized for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Natacha ENTZ-WERLE, MD, PhD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (9):
- France (9):
  - Hôpital des Enfants - Groupe Hospitalier Pellegrin, Bordeaux
  - Centre Oscar Lambret, Lille
  - Institut Hémato-Oncologie Pédiatrique (IHOP), Lyon
  - CHU La Timone, Marseille
  - CHU Mère-Enfants, Nantes
  - Institut Curie, Paris
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Hôpital des Enfants, Toulouse
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Result] Jannier S, Kemmel V, Sebastia Sancho C, Chammas A, Sabo AN, Pencreach E, Farace F, Chenard MP, Lhermitte B, Geoerger B, Aerts I, Frappaz D, Leblond P, Andre N, Ducassou S, Corradini N, Bertozzi AI, Guerin E, Vincent F, Velten M, Entz-Werle N. SFCE-RAPIRI Phase I Study of Rapamycin Plus Irinotecan: A New Way to Target Intra-Tumor Hypoxia in Pediatric Refractory Cancers. Cancers (Basel). 2020 Oct 20;12(10):3051. doi: 10.3390/cancers12103051. PMID 33092063